CLINICAL TRIAL: NCT07238686
Title: Phase 2 Study of Venetoclax-containing Therapy in Combination With HLA-mismatched Mobilized Peripheral Blood Mononuclear Cell Infusion for Intermediate-risk and Higher Myelodysplastic Syndromes
Brief Title: Venetoclax-containing Therapy Combined With Microtransplant for Intermediate-risk and Higher MDS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEN-MST for MDS
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: venetoclax; hypomethylating agent; GPBMC infusion; microtransplant; microtransplantation
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — venetoclax; Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): This cohort includes patients with intermediate-risk and higher MDS who are ineligible for or refuse allogeneic HSCT. Patients receive Venetoclax in combination with hypomethylating agent and HLA-mismatched donor GPBMC infusion. Treatment cycles are 28 days, repeated until disease progression or unacceptable toxicity.
  Interventions: Drug: Venetoclax; Drug: Azacitidine (AZA) or Decitabine (DAC); Biological: GPBMC infusion

INTERVENTIONS:
Drug: Venetoclax — Given PO. For the first cycle, dose of 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Days 3-14. For other cycles, dose of 400 mg on Days 1-14. Note: The dose should be reduced to 100-200 mg daily if concomitant azole antifungals are required.
Drug: Azacitidine (AZA) or Decitabine (DAC) — AZA: Given SC. Dose of 75 mg/m² on Days 1-7 of each cycle. DAC: Given IV. Dose of 20 mg/m² on Days 1-5 of each cycle.
Biological: GPBMC infusion — HLA-mismatched donor GPBMCs are infused on Day 15.

SUMMARY:
This study aims to evaluate the safety and efficacy of a Venetoclax and hypomethylating agent-based regimen combined with infusion of HLA-mismatched donor G-CSF mobilized peripheral blood mononuclear cells (GPBMC) in patients with intermediate-risk and higher myelodysplastic syndromes who are ineligible for allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, male or female, non-limited by race or ethnicity.
* Confirmed diagnosis of MDS according to the World Health Organization (WHO) 5th edition classification, based on histopathology and cytogenetics.
* Risk stratification according to the Revised International Prognostic Scoring System (IPSS-R) must place the patient in the intermediate-, high-, or very high-risk category.
* Not candidates for or refuse allogeneic hematopoietic stem cell transplantation.
* Adequate hepatic function including alanine transaminase (ALT) and aspartate aminotransferase (AST )<= 3 × upper limit of normal(ULN), and total bilirubin <= 1.5 × ULN.
* Adequate renal function including serum creatinine <= 2 × ULN or CrCl>= 40mL/min.
* LVEF measured by echocardiogram is within the normal range (LVEF > 50%).
* The subject must have one donor who is >= 18 years old and HLA matched at 0-7/10 loci (i.e., at least 3 HLA loci must be mismatched). In addition, the donor voluntarily donates hematopoietic stem cells and signs the consent form.
* Each subject (or his/her legal representatives) must sign the Informed Consent Form (ICF), indicating that he/she understands the purpose and procedures of research, and is willing to participate in research.
* Donor inclusion criteria: The donor meets the institution's criteria for related peripheral blood hematopoietic stem cell donors. The donor must be able to tolerate the cell separation and collection process, and sign the Informed Consent Form.

Exclusion Criteria:

* Uncontrolled infection or hemorrhage.
* Cardiovascular disease with clinical significance, such as uncontrolled or highly symptomatic cardiac arrhythmias, congestive heart failure, or myocardial infarction within 6 months prior to screening, or New York Heart Association (NYHA) function class 3 (moderate) or class 4 (severe) heart disease.
* Uncontrolled autoimmune disease or requiring immunosuppression treatment.
* History of severe blood infusion reaction.
* Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception.
* Psychiatric disorder or cognitive impairment that in the researcher's judgment would make the subject not likely to adhere to the protocol requirements.
* Major surgery within 4 weeks prior to enrollment.
* Life-threatening illness other than MDS or uncontrolled intercurrent illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Measured up to 4 years after the last participant is enrolled
  OS is defined as the number of days from the date of study entry to the date of death.
Overall response rate (ORR) | Measured up to 2 years after the last participant is enrolled
  ORR is defined as complete remission (CR) (or CR equivalent) + partial remission (PR) + CR with limited count recovery (CRL) + CR with partial hematologic recovery (CRh) + hematologic improvement (HI) according to IWG 2023 criteria.

SECONDARY OUTCOMES:
Modified overall response (mOR) | Measured up to 2 years after the last participant is enrolled
  Modified OR is defined as CR+PR+CRL+CRh.
Complete remission (CR) | Measured up to 2 years after the last participant is enrolled
  CR is defined as absolute neutrophil count > 1 × 109/L, platelet count > 100 × 109/L, Hb ≥10 g/dL, bone marrow with < 5% blasts, and PB blasts 0%.
Partial remission (PR) | Measured up to 2 years after the last participant is enrolled
  PR is defined as decrease of at least 50% in the percentage of blasts still ≥5% in the bone marrow, peripheral blood neutrophil count > 1 × 109/L, platelet count > 100 × 109/L, Hb ≥10 g/dL.
CR with limited count recovery (CRL) | Measured up to 2 years after the last participant is enrolled
  CRL is defined as bone marrow with less than 5% blasts, PB blasts 0%, and PB only meeting 1 or 2 of the following: absolute neutrophil count > 1 × 109/L, platelet count > 100 × 109/L, Hb ≥10 g/dL.
CR with partial hematologic recovery (CRh) | Measured up to 2 years after the last participant is enrolled
  CRh is defined as bone marrow with less than 5% blasts, and PB not meeting criteria for CR or CRL, no Hb threshold required, platelets ≥50 × 109/L, neutrophils ≥0.5 × 109/L, blasts 0%.
Progression-free survival (PFS) | Measured up to 4 years after the last participant is enrolled
  PFS is defined as the number of days from the date of study entry to the date of the first of the following events: progressed disease; relapse from CR (or CR equivalent), PR, CRL, CRh, or HI; death from any cause.
Treatment-related mortality (TRM) | Measured up to 2 years after the last participant is enrolled
  TRM is defined as the death related to treatment instead of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Cai, MD, Principal Investigator — Department of Hematology, the Fifth Medical Center of Chinese PLA General Hospital
Locations (1):
- Department of Hematology, the Fifth Medical Center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No